CLINICAL TRIAL: NCT06913634
Title: Observational Study to Evaluate the Long- Term Safety and Efficacy of Luspatercept in Subjects Who Received at Least One Dose of Luspatercept in the "Compassionate" Use Phase
Brief Title: Study to Evaluate the Long- Term Safety and Efficacy of Luspatercept in Subjects Who Received at Least One Dose of Luspatercept in the Compassionate Use Phase
Acronym: LUSPA001
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione per la Ricerca sulle Anemie ed Emoglobinopatie in Italia (Other)
Responsible Party: Sponsor
Other Study IDs: LUSPA001
Record Dates: First submitted 2025-02-25; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-02

CONDITIONS: Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia | interventions — luspatercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Luspatercept (ACE-536) — Luspatercept (ACE-536)

SUMMARY:
Luspatercept represents the first and only erythroid maturation agent (EMA) approved by the European Commission (EC) and the Food and Drug Administration (FDA) capable of enhancing advanced erythrocyte maturation.

The efficacy of luspatercept was demonstrated in the phase III clinical trial called "BELIEVE." More than 200 Italian patients with transfusion- dependent beta thalassemia aged ≥18 years who had no approved therapeutic alternatives to improve their clinical course were considered eligible for the 'compassionate' use program related to luspatercept and most of them received at least one dose of the drug before it was dispensed by the National Health System (NHS), after approval by the pharmaceutical company and the Ethics Committee of the Clinical Center in which they were being followed.

DETAILED DESCRIPTION:
One month after the publication in the Official Gazette of the Italian Republic of the AIFA determination of price and reimbursement for the treatment indication covered by the program, those who were still on treatment and were, in clinical judgment, eligible to continue it, continued to receive the drug through dispensation by the NHS.

Because access to the compassionate phase was less restrictive than access to that in formal clinical trials and the patients included particularly representative of real life, collecting data on clinical characteristics at baseline, safety, and efficacy is critical to enriching the information available on this new therapy. Continuing to collect efficacy, safety, and tolerability information beyond the compassionate phase is also essential for a more complete and accurate assessment, given the short duration of 'compassionate' treatment for a portion of the patients under study.

ELIGIBILITY:
Inclusion criteria:

- Subjects who received at least one dose of luspatercept in the compassionate phase

Exclusion Criteria:

- Subjects who are not willing or able to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (male and female), living or deceased patients with transfusion-dependent beta thalassemia who received at least one dose of luspatercept during the compassionate use program.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety of luspatercept, number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12-week interval period of luspatercept treatment.
  To evaluate safety of luspatercept in subjects with transfusion-dependent beta thalassemia who received at least one dose of the drug in the compassionate use phase including the post- marketing authorisation phase in those who continued to receive it.
To evaluate tolerability of luspatercept, number of participants with treatment-related adverse events as assessed by CTCAE v4.0" | 12-week interval period of luspatercept treatment.
  To evaluate tolerability of luspatercept in subjects with transfusion-dependent beta thalassemia who received at least one dose of the drug in the compassionate use phase including the post- marketing authorisation phase in those who continued to receive it.
To evaluate efficacy of luspatercept, Number of subjects who showed a ≥ 33% reduction from baseline in the number of transfused blood units during any 12-week interval period of luspatercept treatment | 12-week interval period of luspatercept treatment.
  To evaluate efficacy of luspatercept in subjects with transfusion-dependent beta thalassemia who received at least one dose of the drug in the compassionate use phase including the post- marketing authorisation phase in those who continued to receive it.

SECONDARY OUTCOMES:
subjects with comorbidities, number of participants with treatment-related adverse events as assessed by CTCAE v4.0" | 12-week interval period of luspatercept treatment.
  To evaluate safety of luspatercept in subjects with comorbidities that were exclusion criteria in formal clinical trials
subjects with comorbidities, number of participants with treatment-related adverse events as assessed by CTCAE v4.0" | 12-week interval period of luspatercept treatment.
  To evaluate tolerability of luspatercept in subjects with comorbidities that were exclusion criteria in formal clinical trials

OTHER OUTCOMES:
endocrinological changes | 52-week interval period of luspatercept treatment.
  Number of subjects who developed endocrinologicalchanges (alterations in frequency and duration of menstrual cycle, alterations in sexual function in men, thyroid dysfunction etc )
thromboembolic events | 52-week interval period of luspatercept treatment.
  New cases of thromboembolic events
factors positively affect drug response | 52-week interval period of luspatercept treatment.
  This outcome will assess the clinical, haematological, and biochemical factors that are positively associated with a favourable drug response to luspatercept, defined as a ≥33% reduction in transfusion burden sustained for at least 12 consecutive weeks during the 52-week treatment period.
  Factors evaluated will include:
  * Baseline haemoglobin level
  * Serum erythropoietin concentration
  * Reticulocyte count
  * Baseline transfusion burden
factors negatively affect drug response | 52-week interval period of luspatercept treatment.
  This outcome will evaluate clinical, haematological, biochemical, or genetic factors that are **associated with a poor or absent response** to luspatercept treatment.
  Non-response will be defined as failure to achieve a ≥33% reduction in transfusion burden for at least 12 consecutive weeks during the 52-week treatment period.
  The following factors will be assessed as potentially associated with a negative response to treatment:
  High baseline transfusion burden Elevated baseline serum erythropoietin levels Lack of reticulocyte increase during treatment Presence of chronic comorbidities (e.g., liver disease, endocrine disorders)
become transfusion independent while taking the drug | 52-week interval period of luspatercept treatment.
  Number of subjects who have not had red blood cell transfusions for at least eight consecutive weeks during treatment

CONTACTS AND LOCATIONS:
Overall Officials: RAFFAELLA ORIGA, Principal Investigator — UNIVERSITA' DI CAGLIARI
Locations (1):
- University of Cagliari, Ospedale Pediatrico Microcitemico, via Jenner sn, 09121 Cagliari -, Cagliari, CA, Italy

IPD SHARING:
Plan to Share IPD: No